CLINICAL TRIAL: NCT02032225
Title: Obtention d'un modèle Cellulaire de la Maladie CADASIL à Partir de Fibroblastes cutanés de Patients
Brief Title: Generation of a Cellular Model of CADASIL From Skin Fibroblasts
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C13-34; 2013-A00994-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-01-03; First posted 2014-01-09 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2016-12

CONDITIONS: CADASIL
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin biopsies will be collected to derive fibroblasts. These will be retained and reprogrammed to iPS cells (also to be retained). iPS cells will be differentiated in vascular smooth muscle cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CADASIL: patients with CADASIL
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy

SUMMARY:
Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leucoencephalopathy (CADASIL) is an archetypal small vessel disease of the brain caused by dominant mutations in the NOTCH3 receptor. Cardinal vascular lesions include deposition of granular osmiophilic material (GOM) within the basal lamina of smooth muscle cells, progressive smooth muscle cell loss, and fibrosis of the media. Pathogenic mutations alter the number of cysteine residues in the extracellular domain of NOTCH3 (Notch3 ECD), leading to its abnormal accumulation in the GOM deposits. Vascular smooth muscle cell has been identified as the primary target cell in this disease. Pathophysiological processes leading from NOTCH3 mutations to smooth muscle cell loss remain poorly understood.

The investigators propose to study these mechanisms by reprogramming skin cells to become stem cells and then differentiating them to vascular smooth muscle cells.

The hypothesis of this study is that the differentiated smooth muscle cells will display the characteristic features of CADASIL, ie, Notch3 ECD accumulation and GOM deposits.

ELIGIBILITY:
Inclusion Criteria :

* Between 30 and 60 years;
* Having a social security scheme or, CMU ;
* Diagnosis of CADASIL confirmed by molecular analysis performed previously (missense mutation in the Notch3 gene affecting the number of cysteine in one of the 34 EGFR of NOTCH3 ) ;
* No countra-indication for a skin biopsy (ongoing treatment with anti-coagulant, history of bleeding disorder or deficiency of blood clotting factors) ;
* Written consent given.

Exclusion Criteria :

* Patients without social security scheme or, CMU ;
* Patients aged under 30 or over 60 years at the time of the first visit ;
* Pregnant women beyond the 5th month of pregnancy
* Patients who are not able to give informed consent ;
* Countra-indication to the achievement of the skin biopsy ( ongoing treatment with anti- coagulant, history of bleeding disorder or deficiency of coagulation factors ) .

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with CADASIL managed at the reference centre for rare vascular diseases of the central nervous system and the retina (CERVCO) (Lariboisière Hospital, Paris, France)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02-11 (Actual); Study Completion 2015-02-11 (Actual)

PRIMARY OUTCOMES:
Derivation of iPS cells from skin biopsies of patients with CADASIL | 30 months

SECONDARY OUTCOMES:
Differentiation of iPS cells to vascular smooth muscle cells, phenotypic and mechanistic analyses | 24 mois
  Differentiation of iPS cells to vascular smooth muscle cells and phenotypic analysis (12 mois) Mechanistic analyses (12 mois)

CONTACTS AND LOCATIONS:
Overall Officials: Anne JOUTEL, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- INSERM, Paris, Paris, France